CLINICAL TRIAL: NCT01746381
Title: Initiation of Long-term Home Non-invasive Ventilation in Amyotrophic Lateral Sclerosis (ALS) Using the iVAPS Mode During a Daytime Trial
Brief Title: Non-invasive Ventilation in Amyotrophic Lateral Sclerosis (ALS) Using the iVAPS Mode
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marta Kaminska (Other)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor-Investigator, Marta Kaminska, Assistant professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2902
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: amyotrophic lateral sclerosis; non-invasive ventilation; home ventilation; IVAPS; neuromuscular diseases
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IVAPS mode of non-invasive ventilation (Experimental): Patients with ALS randomized to this arm will be treated with non-invasive home ventilation using the Intelligent Volume-Assured Pressure Support (IVAPS) mode
  Interventions: Device: Non-invasive home ventilation
- BIST mode of non-invasive ventilation (Active Comparator): Patients with ALS who are randomized to this arm will receive non-invasive home ventilation with the traditional bilevel non-invasive ventilation in spontaneous/timed (BIST) mode
  Interventions: Device: Non-invasive home ventilation

INTERVENTIONS:
Device: Non-invasive home ventilation — A ventilator and mask will be provided to patients according to standard procedures used at the National Program of Home Ventilatory Assistance of the Montreal Chest Institute, adjusted during a daytime outpatient trial, with close follow-up as described in study protocol.
  Other Names: Resmed Stellar 150

SUMMARY:
Home non-invasive ventilation (NIV) is the standard-of-care as initial therapy for patients with ALS with worsening symptoms or deteriorating respiratory function, and has been recommended by the American Academy of Neurology (AAN) practice parameter for ALS.

This study will compare the current standard BiST mode of ventilation with the new iVAPS mode. The main study hypothesis is that the iVAPS mode, initiated in a single daytime trial, will result in a reduction of the number of respiratory therapist interventions and changes in ventilator settings as compared with the standard BiST mode. This will be assessed over a period of one year. In addition this study will test whether the iVAPS mode is superior to BiST mode with respect to: comfort and ease of use; improvement in nighttime and daytime symptoms of hypoventilation; compliance (hours used per day); physiologic parameters (daytime and overnight oxygen saturation and transcutaneous CO2 level).

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disorder that is incurable, progressive, manifested by muscle weakness and wasting, and caused by degeneration of motor neurones. The limited data available suggest the incidence of ALS in Canada to be approximately 2 per 100,000 persons. The disease is characterized by progressive weakness of respiratory muscles, leading to respiratory insufficiency which is often the cause of death in patients with ALS.

Home non-invasive ventilation (NIV) is the standard-of-care as initial therapy for patients with ALS with worsening symptoms or deteriorating respiratory function, and has been recommended by the American Academy of Neurology (AAN) practice parameter for ALS. The symptomatic and survival benefits offered by NIV to patients with ALS make the optimization of ventilation a priority in terms of physiological variables but also symptoms to improve comfort, and consequently, compliance.

The Intelligent Volume-Assured Pressure Support (iVAPS) is a ventilator mode on the Stellar 150 ventilator (Resmed) that uses an algorithm to target alveolar ventilation. It has a learning mode to determine the initial optimal settings to commence ventilation, and is an adaptive mode, which constantly monitors the patient's spontaneous ventilation and adjusts the level of pressure support to maintain target alveolar ventilation.

The aim of the study is to determine the feasibility of long-term non-invasive home ventilation in ALS patients using the Stellar 150 IVAPS mode, initiated during a single daytime trial, and to assess the number of respiratory therapist interventions subsequently required as well as several patient-centered outcomes. The study will be conducted among patients with ALS referred to the National Program of Home Ventilatory Assistance (NPHVA) at the Montreal Chest Institute. The province-wide program provides home ventilation services to patients with a variety of neuromuscular and other disorders. Referred patients will be randomized to receive traditional Bilevel ventilation in ST mode (BiST) or iVAPS and will be followed over a period of one year. Respiratory therapist interventions (beyond scheduled visits) and changes in ventilator settings will be based on patient complaints and aimed at optimizing patient comfort and ventilator use. In addition, symptoms questionnaires will be administered regularly, overnight oxymetry and transcutaneous capnography (at 6 and 12 months) will be performed. Compliance data will be assessed regularly from ventilator memory downloads at each of the scheduled respiratory therapist home visits (1 week, 1, 6 and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the National Program of Home Ventilatory Assistance (NPHVA) at the Montreal Chest Institute for home ventilation.
* Patients that meet eligibility criteria for home ventilation as per the Quebec Health Ministry reference frame document for home ventilation (http://publications.msss.gouv.qc.ca/acrobat/f/documentation/2011/11-936-01W.pdf).
* Adequate knowledge of English or French to complete study questionnaires.

Exclusion Criteria:

* The lack of eligibility for home ventilation, as per the document mentioned above
* Active cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Difference in the number of respiratory therapist interventions required using IVAPS vs BIST mode of ventilation in patients with ALS. | One year
  The investigators define interventions as any complaint from the patient related to the ventilator that warrants an unscheduled visit from the respiratory therapist or a change in ventilator settings.

SECONDARY OUTCOMES:
Feasibility of initiating long term home ventilation in ALS patients using the Stellar 150 iVAPS mode during a single daytime trial. | 1 month
  This will be determined by compliance with use of nocturnal ventilation at 1 month, and good control of nocturnal oxygenation and sleep-disordered breathing at 1 week.
Difference in symptoms with IVAPS vs. BiST in ALS patients | 1,6,12 months
  The investigators will use a questionnaire to assess hypoventilation-related symptoms and comfort with the ventilator.
Effectiveness of ventilation by IVAPS vs. BiST on night-time respiratory parameters in ALS patients | 1 week, 6 months, 12 months
  This will be measured at 1 week using the Embletta portable monitor and transcutaneous capnography, and at 6 and 12 months using overnight oximetry and transcutaneous capnography.
Long-term compliance with the use of nocturnal ventilation on IVAPS vs. BiST in ALS patients | 1,6,12 months
  This will be determined by the number of hours use per day recorded by the device.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Kaminska, MD,MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Rita Troini, RRT,MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Chest Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Radunovic A, Mitsumoto H, Leigh PN. Clinical care of patients with amyotrophic lateral sclerosis. Lancet Neurol. 2007 Oct;6(10):913-25. doi: 10.1016/S1474-4422(07)70244-2. PMID 17884681
- [Background] Piper AJ, Sullivan CE. Effects of long-term nocturnal nasal ventilation on spontaneous breathing during sleep in neuromuscular and chest wall disorders. Eur Respir J. 1996 Jul;9(7):1515-22. doi: 10.1183/09031936.96.09071515. PMID 8836668
- [Background] Aboussouan LS, Khan SU, Meeker DP, Stelmach K, Mitsumoto H. Effect of noninvasive positive-pressure ventilation on survival in amyotrophic lateral sclerosis. Ann Intern Med. 1997 Sep 15;127(6):450-3. doi: 10.7326/0003-4819-127-6-199709150-00006. PMID 9313002
- [Background] Pinto AC, Evangelista T, Carvalho M, Alves MA, Sales Luis ML. Respiratory assistance with a non-invasive ventilator (Bipap) in MND/ALS patients: survival rates in a controlled trial. J Neurol Sci. 1995 May;129 Suppl:19-26. doi: 10.1016/0022-510x(95)00052-4. PMID 7595610
- [Background] McKim DA, Road J, Avendano M, Abdool S, Cote F, Duguid N, Fraser J, Maltais F, Morrison DL, O'Connell C, Petrof BJ, Rimmer K, Skomro R; Canadian Thoracic Society Home Mechanical Ventilation Committee. Home mechanical ventilation: a Canadian Thoracic Society clinical practice guideline. Can Respir J. 2011 Jul-Aug;18(4):197-215. doi: 10.1155/2011/139769. PMID 22059178
- [Background] Atkeson AD, RoyChoudhury A, Harrington-Moroney G, Shah B, Mitsumoto H, Basner RC. Patient-ventilator asynchrony with nocturnal noninvasive ventilation in ALS. Neurology. 2011 Aug 9;77(6):549-55. doi: 10.1212/WNL.0b013e318228c0fb. Epub 2011 Jul 27. PMID 21795658
- See also: Quebec Home Ventilation Program — http://publications.msss.gouv.qc.ca/acrobat/f/documentation/2011/11-936-01W.pdf